CLINICAL TRIAL: NCT05938075
Title: Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of VXCO-100 in Adults in the Republic of South Africa
Brief Title: Study of VXCO-100, a SARS-CoV Candidate Vaccine, in Adults in the Republic of South Africa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaccine Company, Inc. (Industry)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VC 102
Record Dates: First submitted 2023-07-05; First posted 2023-07-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: SARS-CoV; SARS-CoV-2
Keywords: Covid-19; SARS-CoV-2; Coronavirus; Vaccine; Sarbecoviruses; Covid
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Coronavirus Infections | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- VXC0-100 at Dose level 1 (Experimental): Participants will receive VXCO-100 at Dose Level 1 via intramuscular (IM) injection on Day 1 and then an optional boost of VXCO-100 at Dose Level 1 on Month 6.
  Interventions: Biological: VXCO-100
- VXC0-100 at Dose level 2 (Experimental): Participants will receive VXCO-100 at Dose Level 2 via intramuscular (IM) injection on Day 1 and then an optional boost of VXCO-100 at Dose Level 2 on Month 6.
  Interventions: Biological: VXCO-100
- VXC0-100 at Dose level 3 (Experimental): Participants will receive VXCO-100 at Dose Level 3 via intramuscular (IM) injection on Day 1 and then an optional boost of VXCO-100 at Dose Level 3 on Month 6.
  Interventions: Biological: VXCO-100
- COVID-19 mRNA vaccine (Experimental): Participants will receive a COVID-19 mRNA vaccine on Day 1 and then a boost with the same COVID-19 mRNA vaccine at Day 21.
  Interventions: Biological: COVID-19 mRNA vaccine

INTERVENTIONS:
Biological: VXCO-100 — Sterile suspension for injection
  Arms: VXC0-100 at Dose level 1; VXC0-100 at Dose level 2; VXC0-100 at Dose level 3
Biological: COVID-19 mRNA vaccine — Sterile suspension for injection
  Arms: COVID-19 mRNA vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of ascending dose levels of VXCO-100 in adults.

DETAILED DESCRIPTION:
This is a phase 1, multisite clinical trial to evaluate the safety and immunogenicity of 3 dose levels of VXCO-100 in adults.

Participants will be vaccinated with a selected dose of VXCO-100 or a COVID-19 mRNA vaccine. Participants will receive a dose of VXCO-100 on Day 1. A matched optional boost on month 6 will be offered to a subset of participants in Groups 1-3. Participants receiving a COVID-19 mRNA vaccine will be vaccinated on Day 1 and Day 21.

Safety will be evaluated before proceeding to a higher dose level.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all the following criteria to be eligible for the study:

1. Adults ages 18 years and older
2. Judged by the investigator to be healthy based on participant-reported medical history, physical examination, vital signs, and laboratory assessment.
3. Able to provide written informed consent.
4. Willing to disclose prior COVID-19 vaccination status.
5. Willing to disclose prior participant-reported SARS-CoV-2 infection status.
6. Willing to comply with all study procedures during the follow-up period of approximately 12 months.
7. Body mass index of ≤ 40 kg/m2 within 30 days prior to enrollment
8. Electrocardiogram (ECG) without clinically significant abnormalities.
9. Clinical screening laboratory evaluations (i.e., CBC, iron, ferritin, TIBC, platelets, ALT, AST, creatinine) are within acceptable normal reference ranges at the clinical laboratory being used or are not deemed clinically significant by study clinician.

   For participants of childbearing potential:
10. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on the day of enrollment
11. Must agree to avoid pregnancy from 21 days prior to study Day 1 until at least 90 days after last study vaccination.

Exclusion Criteria:

A participant will be excluded if one or more of the following conditions apply:

1. Known SARS-CoV-2 infection or positive test result within 6 months prior to Day 1
2. Ongoing prophylactic COVID-19 treatment, or monoclonal antibody infusion within 6 months prior to Day 1
3. Any COVID-19 vaccination within 6 months prior to Day 1
4. Exhibits symptoms consistent with COVID-19 as assessed by study clinician such as: fever, dry cough, fatigue, nasal obstruction, runny nose, sore throat, myalgia, diarrhea, shortness of breath or dyspnea within 14 days prior to in Day 1
5. Known close contact (as defined by CDC, 2021a) with someone who has COVID-19 within 14 days prior to Day 1
6. History or presence of self-reported or medically documented significant medical or psychiatric condition(s) as assessed by study clinician, including:

   1. At high risk of severe COVID-19 disease, such as significant history of COPD or chronic lung disease, chronic kidney disease, serious heart conditions (such as heart failure, coronary artery disease or cardiomyopathies), sickle cell disease, diabetes
   2. Clinically significant central nervous system disease such as epilepsy, encephalopathy, or a history of severe mental illness
   3. Severe liver and/or kidney diseases, uncontrolled hypertension, or ongoing or highly likely to recur malignancies
   4. Ongoing or recent clinically significant history of alcohol or drug abuse
7. Active participation in an interventional clinical study with an investigational drug/biologic/device agent receipt of any specimen collection within 30 days prior to Day 1
8. Evidence of infection with hepatitis B virus or hepatitis C virus
9. Positive test result for human immunodeficiency virus (HIV) with the exception that 30% of participants may be HIV-infected, if stable on antiretrovirals with stable CD4 >350 cells/mm3 and virally suppressed
10. History of myocarditis or pericarditis
11. Diagnosed with congenital or acquired immune deficiency, ongoing lymphoma, leukemia, or other clinically significant immune compromising or autoimmune conditions.
12. History of known coagulation dysfunction (e.g., coagulation factor deficiency, known thrombocytopenia, platelet dysfunction, coagulation disease, etc.)
13. Receipt of any live attenuated vaccine within 30 days, or with any other (non-live) vaccine within 14 days prior to Day 1
14. Received more than 10 days of any systemic immunosuppressants or cytotoxic medications within 30 days prior to Day 1, any within 14 days prior to Day 1 or is anticipating the need for immunosuppressants at any time during participation in the study.
15. Received any blood products within 3 months prior to Day 1
16. Donated > 450 mL of whole blood within 30 days prior to Day 1
17. History of unexplained or recurrent anaphylaxis or angioedema, or a history of severe allergic reaction (e.g., anaphylaxis) after a previous dose of any vaccine, or to any component of VXCO-100.
18. For persons of childbearing potential: breastfeeding or planning to become pregnant during trial duration.
19. Any condition that, in the opinion of the investigator, would (a) pose a health risk to the participant if enrolled or (b) could interfere with evaluation of the study vaccine or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with solicited local adverse events | For 7 days after each product administration
Number and percentage of participants with solicited systemic adverse events | For 7 days after each product administration
Number and percentage of participants with unsolicited and safety laboratory-based adverse events | For 28 days after each product administration
Numbers and percentages of participants with serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs), medically attended adverse events (MAAEs), and adverse events of special interest (AESIs) | For 364 days after each product administration

SECONDARY OUTCOMES:
Response rate measured by geometric mean titer of the serum neutralizing antibody (Nab) against the ancestral (Wuhan) strain | At baseline and 21 days after each product administration
Response rate measured by GMT of Nab against selected variants of concern | At baseline and 21 days after each product administration
Numbers and percentages of participants with positive Th1 or Th2 cytokine responses for CD4 and CD8 as measured by multi-parameter intracellular cytokine staining | At baseline and 7 days after each product administration

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Gray, MBChB, FC, Principal Investigator — Medical Research Council, South Africa; Ravindre Panchia, MBChB, Principal Investigator — Perinatal HIV Research Unit (PHRU); Anusha Nana, BPharm, Principal Investigator — Perinatal HIV Research Unit (PHRU); Mbalizethu Mntambo, MBChB, Principal Investigator — HIV and other Infectious Diseases Research Unit (HIDRU); Samantha Siva, MMEDSc, Principal Investigator — HIV and other Infectious Diseases Research Unit (HIDRU)
Locations (2):
- South Africa (2):
  - Perinatal HIV Research Unit (PHRU), Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng
  - HIV and other Infectious Diseases Research Unit (HIDRU), South African Medical Research Council, Botha’s Hill, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: No